CLINICAL TRIAL: NCT00927069
Title: Open Label Study to Evaluate the Efficacy and Safety of Adalimumab in Patients With Plaque Psoriasis Who Showed an Unsatisfactory Response to Etanercept
Brief Title: Safety and Efficacy of Adalimumab in Patients Who Showed an Unsatisfactory Response to Etanercept
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innovaderm Research Inc. (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Inno-6002
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Results first posted 2010-08-24 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Plaque Psoriasis
Keywords: Adalimumab
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Experimental): Patients who have shown an unsatisfactory response to 3 months of etanercept 50 mg twice a week without dose reduction prior to screening.
  Interventions: Drug: Adalimumab every other week
- Group B (Experimental): Patients who showed a satisfactory response to 3 months or more of etanercept 50 mg twice a week followed by a loss of response after dose reduction to 50 mg etanercept once a week prior to screening.
  Interventions: Drug: Adalimumab every other week
- Group A dose increase at Week 12 (Experimental): Patients in group A who - after 12 weeks of adalimimab 40 mg every other week in this study - failed to reach a physician's global assessment (PGA) of clear or almost clear and had a dose increase to 40 mg adalimimab every week for another 12 weeks.
  Interventions: Drug: Adalimumab Every Week
- Group B dose increase at Week 12 (Experimental): Patients in group B who - after 12 weeks of adalimimab 40 mg every other week in this study - failed to reach a physician's global assessment (PGA) of clear or almost clear and had a dose increase to 40 mg adalimimab every week for another 12 weeks.
  Interventions: Drug: Adalimumab Every Week

INTERVENTIONS:
Drug: Adalimumab every other week — Adalimumab 40mg injection every other week for 24 weeks
  Other Names: HUMIRA
  Arms: Group A; Group B
Drug: Adalimumab Every Week — Adalimumab 40mg injection every week for the last 12 weeks of study.
  Other Names: HUMIRA
  Arms: Group A dose increase at Week 12; Group B dose increase at Week 12

SUMMARY:
This study will provide data on additional therapeutic benefits in administering Adalimumab in patients with plaque psoriasis that showed an unsatisfactory response after at least 3 months of treatment with etanercept.

DETAILED DESCRIPTION:
A total of 50 patients with psoriasis vulgaris who showed an unsatisfactory response to etanercept 50 mg twice a week followed by 50 mg once a week and a total of 50 patients who showed an unsatisfactory response to etanercept 50 mg twice a week without dose reduction will be recruited. All patients will receive adalimumab 40 mg every other week (EOW) for 12 weeks. Patients who fail to reach a physician's global assessment (PGA) of clear or almost clear at week 12 will have an increase in adalimumab to 40 mg every week (EW) for an additional 12 weeks. Patients who reach a PGA of clear or almost clear at week 12 will continue to receive adalimumab at 40 mg EOW for an additional 12 weeks. Patients will be evaluated for safety and efficacy every 4 weeks for a total of 24 weeks. PASI, BSA and PGA will be performed at each visit. Routine chemistry, hematology and urinalysis will be performed every 4 weeks.

The percentage of patients achieving a physician's global assessment (PGA) of clear or almost clear after at least 12 weeks of adalimumab will be calculated for patients who had shown an unsatisfactory response to 3 months of etanercept at 50 mg twice a week without dose reduction as well as for patients who had shown an unsatisfactory response to 3 months of etanercept at 50 mg twice a week followed by 50 mg once a week.

A physician's global assessment (PGA) of clear is defined by no plaque elevation over normal skin. There is no scale. Erythema is perceptible as hyperpigmentation, pigmented macules, diffuse faint pink or red coloration.

A physician's global assessment (PGA) of almost clear is defined as follows: It is possible but difficilt to ascertain whether there is a slight elevation above normal skin. There is scaling in the form of surface dryness with some white coloration. Erythema is up to a definite red coloration.

ELIGIBILITY:
Inclusion Criteria:

* Subject with plaque psoriasis with documentation of an unsatisfactory response to etanercept as defined by either:

  1. Failure to present a PGA of clear or almost clear after at least 3 months of etanercept at 50 mg twice a week OR;
  2. Failure to present a PGA of clear or almost clear after at least 3 months of etanercept at 50 mg twice a week followed by a dose reduction to 50 mg once a week. To be eligible these patients must have reached a PGA of clear or almost clear after at least 3 months of etanercept at 50 mg twice a week followed by a loss of PGA of clear or almost clear at anytime after a dose reduction to 50 mg of etanercept once a week.
* Subject presents a PGA of 3 or more at baseline visit.
* Subject with plaque psoriasis at screening that is severe enough to be candidate for systemic therapy.
* Subject is 18 to 80 years of age .
* Female subject is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or is of childbearing potential and practicing one of the following methods of birth control throughout the study and for 150 days after study completion:

  1. condoms, sponge, foams, jellies, diaphragm or IUD;
  2. contraceptives (oral or parenteral) for three months prior to study drug administration;
  3. a vasectomized partner;
* Female subjects of childbearing potential must have a negative serum pregnancy test at the Screening visit.
* Subject is judged to be in good general health as determined by the principal investigator based upon the results of medical history, laboratory profile, physical examination, and CXR performed at Screening.
* Subjects will be evaluated for latent TB infection with a PPD test and CHX. Subjects who demonstrate evidence of latent TB infection (either PPD more than or equal to 5 mm of induration, irrespective of BCG vaccination status and negative CXR findings for active TB, and/or suspicious CXR findings will not be allowed to participate in the study.
* Subjects must be able and willing to provide written informed consent and comply with the requirements of this study protocol.
* Subjects must be able and willing to self-administer SC injections or have a qualified person available to administer SC injections.

Exclusion Criteria:

* Subject has other active skin diseases or skin infections (bacterial, fungal, or viral) that may interfere with evaluation of psoriasis or with subject's safety.
* Subject has a history of an allergic reaction or significant sensitivity to constituents of study drug, including latex (a component of the pre-filled syringe).
* Subject who has used topical treatments in the last 4 weeks of the etanercept treatment period when the response to etanercept was evaluated as unsatisfactory must use the same topical therapy with the same agents applied in the same manner and with the same application frequency for two weeks prior to the baseline visit as well as during the entire trial. The use of any other topical treatment for psoriasis is prohibited except for allowed treatments.
* Subject who has used UVB phototherapy, excessive sun exposure, phototherapy or any non-biological systemic therapy for the treatment of psoriasis less than 30 days before day 0. Investigational chemical agents must be discontinued at least 30 days or 5 half-lives prior to the Baseline visit (whichever is longer).
* Subject who has used any biological therapy (apart from etanercept) for the treatment of psoriasis less than 3 months (90 days) before day 0. Etanercept must be discontinued before baseline but a washout period is not required.
* Subject is taking or requires oral or injectable corticosteroids during the study. Inhaled corticosteroids for stable medical conditions are allowed.
* Subjects for whom documentation of unsatisfactory response to etanercept was obtained while the subject was under combination treatment with any of the following: UVB phototherapy, PUVA therapy, prednisone, methotrexate, acitretin, cyclosporine or any other systemic or biologic drug (apart from etanercept).
* Subject has a poorly controlled medical condition, such as uncontrolled diabetes with documented history of recurrent infections, unstable ischemic heart disease, congestive heart failure, recent stroke and any other condition which, in the opinion of the investigator, would put the subject at risk if participating in the study.
* Subject has history of neurologic symptoms suggestive of central nervous system (CNS) demyelinating disease.
* Subject has history of cancer or lymphoproliferative disease other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix.
* Subject has a history of listeriosis, treated or untreated TB, persistent chronic infections, or recent active infections requiring hospitalization or treatment with intravenous anti-infectives within 30 days or oral anti-infectives within 14 days prior to the Baseline visit.
* Subject who has received any live attenuated vaccine 28 days or less before baseline.
* Subject with hepatitis B or hepatitis C viral infection.
* Subject with any of the following: hemoglobin ≤ 10 g/L, white blood cells ≤ 3.0 X 109/L, platelet counts ≤130 X 109/L, ALT ≥ 2 times the upper limit of normal, AST ≥ 2 times the upper normal limit, total bilirubin ≥ 2 times the upper normal limit or creatinine ≥ 150 mmol/L.
* Subject currently uses or plans to use anti-retroviral therapy at any time during the study.
* Subject is known to have immune deficiency or is immunocompromised.
* Female subject who is pregnant or breast-feeding or considering becoming pregnant during the study or for 150 days after the last dose of study medication.
* Subject has a history of clinically significant drug or alcohol abuse in the last year.
* Subject is considered by the investigator, for any reason, to be an unsuitable candidate for the study.
* Subject has erythrodermic psoriasis, generalized or localized pustular psoriasis, medication-induced or medication-exacerbated psoriasis, or new onset guttate psoriasis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2007-03; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Innovaderm Research Inc.
Locations (12):
- Canada (12):
  - Winnipeg Clinic, Winnipeg, Manitoba
  - NewLab Clinical Research, St. John's, Newfoundland and Labrador
  - Mediprobe Research, London, Ontario
  - The Guenther Dermatology Research center, London, Ontario
  - Lynderm Research, Markham, Ontario
  - Entralogix Inc., Oakville, Ontario
  - Entralogix Clinical Group Inc., Toronto, Ontario
  - Windsor Clinical Research Inc., Windsor, Ontario
  - Innovaderm Research Laval Inc., Laval, Quebec
  - Innovaderm Research Inc, Montreal, Quebec
  - Centre de Recherche Clinique Martin Gilbert inc et Centre Dermatologie Maizerets, Québec, Quebec
  - Centre de Recherches Dermatologiques du Quebec Metropolitain, Ste-Foy, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Patients who have shown an unsatisfactory response to 3 months of etanercept wihout dose reduction prior to screening.
- Groupe A Dose Increase at Week 12: Patients in group A who - after 12 weeks of adalimimab 40 mg every other week in this study - failed to acheive a PGA of clear or almost clear and had a dose increase to 40 mg adalimimab every week for another 12 weeks.
- Groupe B Dose Increase at Week 12: Patients in group B who - after 12 weeks of adalimimab 40 mg every other week in this study - failed to acheive a PGA of clear or almost clear and had a dose increase to 40 mg adalimimab every week for another 12 weeks.
Period: Week 0 to Week 12
Arm/Group | Group A | Group B | Groupe A Dose Increase at Week 12 | Groupe B Dose Increase at Week 12
Started | 50 | 35 | 0 | 0
Completed | 49 | 34 | 0 | 0
Not Completed | 1 | 1 | 0 | 0
Not completed — Worsening of psoriasis | 1 | 1 | 0 | 0
Period: Week 12 to Week 24
Arm/Group | Group A | Group B | Groupe A Dose Increase at Week 12 | Groupe B Dose Increase at Week 12
Started | 18 (17 patients stayed at the same dose. One patient withdrew at Week 12 and also had no dose increase) | 11 (11 patients stayed at the same dose of 40 mg Adalimumab every other week) | 31 (31 Pts. from Group A had a dose incr. since they did not respond to 40mg adalimumab every other week) | 23 (23 Pts. from Group B had a dose incr. since they did not respond to 40mg adalimumab every other week)
Completed | 16 | 11 | 28 | 20
Not Completed | 2 | 0 | 3 | 3
Not completed — Lack of Efficacy | 0 | 0 | 2 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Had a vaccination, removed from study | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 50 | 35 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 32 | 79
  >=65 years | 3 | 3 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 49.12 (11.18) | 46.17 (11.2) | 47.91 (11.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 36 | 24 | 60
Region of Enrollment [Number; unit: participants]
  Canada | 50 | 35 | 85

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients From Group B Who Achieve a Physician's Global Assessment (PGA) of Clear or Almost Clear at Week 12.
Description: Efficacy of adalimumab 40 mg every other week in patients in Group B by calculating the number of patients who achieve a PGA of clear or almost clear at Week 12.
  Clear is defined by no plaque elevation above normal skin. There is no scale. Erythema is perceptible as hyperpigmentation, pigmented macules, diffuse faint pink or red coloration.
  Almost Clear is defined as follows: It is possible but difficult to ascertain whether there is a slight elevation above normal skin. There is scaling in the form of surface dryness with some white coloration. Erythema is up to a difinite red coloration.
Time Frame: 12 weeks
Population: The analysis was intent to treat (ITT) and inputed Last observation carried forward (LOCF)
Measure: Number; unit: Participants
Arm/Group | Group B
Number analyzed (Participants) | 35
Participants | 11

2. Secondary Outcome: Number of Patients From Group A Who Achieve a Physician's Global Assessment (PGA) of Clear or Almost Clear at Week 12.
Description: Efficacy of adalimumab in patients from Group A who achieve a Physician's Global Assessment (PGA) of clear or almost clear at week 12.
  Clear is defined by no plaque elevation above normal skin. There is no scale. Erythema is perceptible as hyperpigmentation, pigmented macules, diffuse faint pink or red coloration.
  Almost Clear is defined as follows: It is possible but difficult to ascertain whether there is a slight elevation above normal skin. There is scaling in the form of surface dryness with some white coloration. Erythema is up to a difinite red coloration.
Time Frame: 12 weeks
Population: The analysis was intent to treat (ITT) and inputed Last observation carried forward (LOCF)
Measure: Number; unit: Participants
Arm/Group | Group A
Number analyzed (Participants) | 50
Participants | 17

3. Secondary Outcome: Number of Patients From Group B Who Achieve a Physician's Global Assessment (PGA) of Clear or Almost Clear at Week 24 After a Dose Increase to 40mg Adalimumab Every Week.
Description: Efficacy of adalimumab in patients from Group B who achieve a Physician's global assessment (PGA) of clear or almost clear at Week 24.
  Clear is defined by no plaque elevation above normal skin. There is no scale. Erythema is perceptible as hyperpigmentation, pigmented macules, diffuse faint pink or red coloration.
  Almost Clear is defined as follows: It is possible but difficult to ascertain whether there is a slight elevation above normal skin. There is scaling in the form of surface dryness with some white coloration. Erythema is up to a difinite red coloration.
Time Frame: 24 weeks
Population: The analysis was intent to treat (ITT) and inputed Last observation carried forward (LOCF)
Measure: Number; unit: Participants
Arm/Group | Groupe B Dose Increase at Week 12
Number analyzed (Participants) | 23
Participants | 7

4. Secondary Outcome: Number of Patients From Group A Who Achieve a Physician's Global Assessment (PGA) of Clear or Almost Clear at Week 24 After a Dose Increase to 40mg Adalimumab Every Week.
Description: Efficacy of adalimumab in patients from Group A who achieve a Physician's Global Assessment (PGA) of clear or almost clear at Week 24.
  Clear is defined by no plaque elevation above normal skin. There is no scale. Erythema is perceptible as hyperpigmentation, pigmented macules, diffuse faint pink or red coloration.
  Almost Clear is defined as follows: It is possible but difficult to ascertain whether there is a slight elevation above normal skin. There is scaling in the form of surface dryness with some white coloration. Erythema is up to a difinite red coloration.
Time Frame: 24 weeks
Population: The analysis was intent to treat (ITT) and inputed Last observation carried forward (LOCF)
Measure: Number; unit: Participants
Arm/Group | Groupe A Dose Increase at Week 12
Number analyzed (Participants) | 31
Participants | 10

5. Secondary Outcome: Total Number of Adverse Events for All Patients in the Study.
Description: Safety of adalimumab in patients with plaque psoriasis that showed an unsatisfactory response after at least 3 months of therapy with etanercept
Time Frame: 24 weeks
Population: The analysis was intent to treat (ITT) and inputed Last observation carried forward (LOCF)
Measure: Number; unit: Adverse events
Groups:
- Group A: Patients at screening had shown an unsastifactory response after 3 months of etanercept 50mg twice a week.
- Group B: Patients at screening had shown a satisfactory response to etanercept 50mg twice a week followed by a loss of response after dose reduction to 50mg etanercept once a week.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 50 | 35
Adverse events | 91 | 63

ADVERSE EVENTS:
Time Frame: The period in which adverse events were recorded was between the signing of the informed consent at screening and Week 28 (approximately 32 weeks).
Arm/Group | Group A | Group B
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/35
Other Adverse Events (participants affected / at risk) | 20/50 | 8/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=50) | Group B (N=35)
Common Cold (Infections and infestations) | 4 (5) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 4 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 9 (12) | 2 (3)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (7) | 0 (0)

LIMITATIONS AND CAVEATS:
This was an open label uncontrolled study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less